CLINICAL TRIAL: NCT01120626
Title: Augmentation of the Cholinergic System in Fragile X Syndrome: A Double-Blind Placebo-Controlled Randomized Study of Donepezil
Brief Title: Randomized Controlled Study of Donepezil in Fragile X Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Autism Speaks (Other)
Responsible Party: Principal Investigator, Allan Reiss, Principle Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SU-02042010-4923; Autism Speaks 5907 (Other Grant/Funding Number: Autism Speaks 5907); R34MH085899-01A1 (NIH); SPO#42922 (Other: Stanford University Research Management Group); SPO#45612 (Other: Stanford University Research Management Group); eProtocol 13773 (SQL 96239) (Other: Stanford University IRB)
Record Dates: First submitted 2010-05-07; First posted 2010-05-11 (Estimated); Results first posted 2016-03-17 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-02

CONDITIONS: Fragile X Syndrome
MeSH Terms: conditions — Fragile X Syndrome | interventions — Donepezil; Sugars; Lactose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- donepezil (Active Comparator): donepezil (2.5 mg to 10.0 mg per day for 12 weeks)
  Interventions: Drug: donepezil
- sugar pill (Placebo Comparator): sugar pill (2.5 mg to 10.0 mg per day for 12 weeks)
  Interventions: Drug: sugar pill

INTERVENTIONS:
Drug: donepezil — donepezil (2.5 mg to 10.0 mg per day for 12 weeks)
  Other Names: Aricept
  Arms: donepezil
Drug: sugar pill — sugar pill (2.5 mg to 10.0 mg per day for 12 weeks)
  Other Names: lactose
  Arms: sugar pill

SUMMARY:
Fragile X syndrome (FraX) is the most common known heritable cause of human intellectual disability. Though recent research has revealed much about the genetic and neurobiological bases of FraX, knowledge about specific and effective treatments for affected individuals is lacking. Based on information from both human and animal studies, one cause of intellectual disability in FraX may be related to deficits in a particular brain neurotransmitter system (the "cholinergic" system). Thus, the investigators propose to use a specific medication, donepezil, to augment cholinergic system in adolescents affected by FraX. If found to be effective, the knowledge generated by this research may also be relevant to other developmental disorders that share common disease pathways with FraX.

DETAILED DESCRIPTION:
Fragile X syndrome (FraX), a neurodevelopmental disorder caused by mutations of the FMR1 gene, is the most common known heritable cause of cognitive and behavioral disability in humans. Though research progress pertaining to FraX has been extraordinary in many areas, many critical gaps in knowledge remain. In particular, there is a dearth of information on treatments designed to address the often-serious cognitive and behavioral symptoms of FraX. Like many other developmental disorders, descriptions of treatments for FraX that do exist in the literature are primarily derived from uncontrolled case studies or series, with both pharmacological and behavioral interventions targeted to symptoms associated with phenomenologically defined "co-morbid" diagnoses such as AD/HD, autism spectrum disorders (ASD) or anxiety disorders. These circumstances are suboptimal as such symptom-based treatments represent a low level of specificity with respect to the underlying pathogenesis of cognitive and behavioral problems. Accordingly, new research to develop more effective, disease-specific treatments for persons with FraX is greatly needed.

Converging evidence from our research group and others strongly support a hypothesis of functional cholinergic deficits contributing to cognitive-behavioral dysfunction in FraX. This evidence includes: (1) abnormalities of cholinergic pathway function and neurochemistry observed with functional MRI and 1H-MRS, respectively, in FraX, (2) an analysis of FMR1 expression during human fetal development indicating particularly high expression in cholinergic brain regions, (3) cholinergic system abnormalities detected in the mouse and fly models of FraX, (4) an analysis of the specific profile of cognitive and behavioral deficits in FraX in relation to current knowledge of cholinergic system functions, and, (5) significant improvements in cognition and behavior observed in 12 individuals with FraX during an open-label trial of donepezil, a cholinesterase inhibitor. Accordingly, the proposed project will consist of a double blind, placebo controlled trial of donepezil in 50 individuals with FraX, ages 12 to 29 years. The primary hypothesis is that subjects receiving donepezil will show greater improvements in specific measures of behavior and cognition, relative to the placebo group. In addition to direct benefit to persons affected by FraX, findings from the proposed research are likely to be highly relevant to subgroups of (currently) idiopathic developmental disorders, such as autism, that might share common pathophysiological mechanisms of disease with FraX. Such shared mechanisms could occur through intersecting pathways involving FMR1 protein function or as a result of similarities in the contribution of cholinergic dysfunction to cognitive and behavioral disability.

ELIGIBILITY:
Inclusion Criteria:

1. confirmed genetic diagnosis of fragile X syndrome
2. age >=12, <=29
3. Verbal IQ >= 50, <=75
4. Tanner pubertal stage >= 3

Exclusion Criteria:

1. Current or lifetime DSM-IV diagnosis of bipolar disorder, schizophrenia, schizoaffective disorder, or psychotic disorder, NOS based upon reported history
2. Poorly controlled seizure disorder or taking more than one anticonvulsant (subjects cannot be prescribed carbamazepine, phenytoin, or phenobarbital due to potential interaction effects with donepezil). The investigators will permit one anticonvulsant as monotherapy for seizures if the seizure disorder is well controlled with no evidence of break through seizures within the past year
3. Concomitant or anticipated use of other medications having prominent effects on the cholinergic system (e.g., bethanechol, benztropine, atropine, succinylcholine)
4. Medications or nutritional supplements that have the potential to significantly alter donepezil levels, clinical effects or adverse reactions (antifungal agents, corticosteroids, erythromycin, beta-blockers, calcium channel blockers, NSAIDs, gingko biloba, St. John's wort)
5. Medical illnesses where donepezil could worsen the condition such as asthma, cardiac conduction abnormalities, urinary obstruction or gastrointestinal disease with gastric bleeding
6. Pregnancy or sexually active females not using a reliable method of contraception
7. If considering participation in brain MRI part of the study, then any contraindications for MRI (e.g., orthodontia, metal in or on the body, etc.)

Ages: 12 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2009-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allan L Reiss, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Center for Interdisciplinary Brain Sciences Research at Stanford — http://cibsr.stanford.edu

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 45 participants consented/enrolled in study. Of these, 3 failed to meet inclusion criteria at the baseline visit and thus were not randomized to receive study drug.
Period: Overall Study
Arm/Group | Donepezil | Sugar Pill
Started | 20 | 22
Completed | 19 | 22
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Donepezil | Sugar Pill | Total
Number analyzed (Participants) | 20 | 22 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10 | 9 | 19
  Between 18 and 65 years | 10 | 13 | 23
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 13 | 14 | 27
Region of Enrollment [Number; unit: participants]
  United States | 20 | 22 | 42
Contingency Naming Test (CNT) Performance Score [Mean (Standard Deviation); unit: correct responses per minute] — Baseline Contingency Naming Test (CNT) performance score on Rule 2 (naming shapes) and on Rule 3 (If the inside shape matches the outside shape, name the color, otherwise, name the outside shape). Performance score is the number of correct responses per minute, calculated by dividing the number of correct responses by the time taken to complete the 27 items, and multiplying by 60.
  correct responses per minute
    CNT Performance Rule 2 | 52.63 (18.54) | 38.77 (26.49) | 45.37 (23.83)
    CNT Performance Rule 3 | 23.08 (12.56) | 13.77 (13.44) | 18.21 (13.71)
Aberrant Behavior Checklist (ABC) [Mean (Standard Deviation); unit: units on a scale] — The Aberrant Behavior Checklist is a 58-item symptom checklist for assessing problem behaviors. The ABC was rated by each participant's parent. Each item is rated on a four-point Likert scale ranging from 0 (not at all a problem) to 3 (the problem is severe in degree). The ABC Total score (range 0-174) is the sum of all individual item scores. Higher score indicates more maladaptive behaviors/worse outcome.
  units on a scale | 19.70 (15.34) | 30.77 (25.54) | 21.26 (19.50)

OUTCOME MEASURES:

1. Primary Outcome: Contingency Naming Test (CNT) Performance Score
Description: Week 12 Contingency Naming Test (CNT) performance score on Rule 2 (naming shapes) and on Rule 3 (If the inside shape matches the outside shape, name the color, otherwise, name the outside shape). Performance score is the number of correct responses per minute, calculated by dividing the number of correct responses by the time taken to complete the 27 items, and multiplying by 60. Higher scores indicate faster and more accurate responding.
Time Frame: Week 12
Population: 41 of 42 randomized participants completed the 12-week randomized controlled trial. 37 of 42 randomized participants completed CNT Rule 2 at week 12. 34 of 42 randomized participants completed CNT Rule 3 at week 12.
Measure: Mean (Standard Deviation); unit: correct responses per minute
Arm/Group | Donepezil | Sugar Pill
Number analyzed (Participants) | 19 | 18
correct responses per minute
  CNT Performance Score Rule 2 | 37.05 (14.60) | 40.50 (31.11)
  CNT Performance Score Rule 3 | 66.94 (46.92) | 61.56 (23.06)

2. Secondary Outcome: Aberrant Behavior Checklist (ABC)
Description: The Aberrant Behavior Checklist is a 58-item symptom checklist for assessing problem behaviors. The ABC was rated by each participant's parent. Each item is rated on a four-point Likert scale ranging from 0 (not at all a problem) to 3 (the problem is severe in degree). The ABC Total score (range 0-174) is the sum of all individual item scores. Higher score indicates more maladaptive behaviors/worse outcome.
Time Frame: Week 12
Population: 41 of 42 randomized participants completed the 12-week randomized controlled trial. 39 of 42 participants were administered the ABC at week 12.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Donepezil | Sugar Pill
Number analyzed (Participants) | 18 | 21
units on a scale | 17.56 (13.65) | 24.43 (23.27)

ADVERSE EVENTS:
Arm/Group | Donepezil | Sugar Pill
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/22
Other Adverse Events (participants affected / at risk) | 0/20 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No